CLINICAL TRIAL: NCT04740268
Title: Clinical Trial Study for the Use of Straberi Microneedling Device to Treat Atrophic Acne Scarring
Brief Title: Straberi Microneedling For Atrophic Acne
Acronym: SAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universal Skincare Institute (Other)
Collaborators: Lavish Beauty (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1114
Record Dates: First submitted 2020-09-13; First posted 2021-02-05 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-01

CONDITIONS: Atrophic Acne Scar
Keywords: microneedling; atrophic acne; epistamp; universal skincare institute
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Participants in the Straberi microneedling trial are those who are seeking improvement for atrophic acne scaring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patiant without treatment (Other): Non-Randomized patients with atrophic acne skin conditions
  Interventions: Device: Straberi
- Straberi Microneedling Treatment (Other): Non-Randomized treatment for patients with atrophic acne skin conditions using the Straberi Microneedling device.
  Interventions: Device: Straberi

INTERVENTIONS:
Device: Straberi — The patient's entire face will be treated with the Straberi microneedling devise.
  The following settings will be used as a treatment protocol. Needle length between .02- 1.55 mm
  Other Names: microneedling

SUMMARY:
This pilot study will expand knowledge and application needling using the Straberi microneedling device for the improvement of Atrophic Acne Scarring

DETAILED DESCRIPTION:
This pilot study will expand the knowledge and application of needling using the Straberi microneedling device and its safety and benefits for improving the appearance of atrophic acne scarring. The pilot aims to objectively measure skin quality using the Derma Scan, photographs, and provide objective data showing improvement by way of the Goodman and Barons quantitative scar scale.

ELIGIBILITY:
Inclusion Criteria:

* Derma Scan showing aging including skin texture, wrinkles, brown spots, and pores.
* Patients willing to sign informed consent.
* Patients willing to be photographed and video documented
* Patients willing to consent to 3 months of treatment

Exclusion Criteria:

* History of eczema in the treatment area; psoriasis and any other chronic skin conditions
* History of actinic (solar) keratosis in the treatment area;
* History of hemophilia
* History of diabetes
* The presence of raised moles, warts on the targeted area.
* Collagen vascular diseases or cardiac abnormalities
* Blood clotting problems
* Active bacterial or fungal infection
* Facial melanosis
* Malignant tumors
* Immunosuppression
* Use of blood thinners or prednisone
* Corticosteroids within two weeks of the procedure
* Chronic liver disease
* Porphyria or other skin diseases.
* Patient not willing to sign informed consent.
* TCA peels in the last 5 weeks
* Subject currently has moderate to severe acne on the face.
* Microneedling within the last 6 months
* Subject has an active infection.
* Subject has a history of a bleeding disorder
* Subject has a history of keloidal tendency
* Subject has received ablative or non-ablative laser treatments in the previous 6 months.
* Subject has taken Accutane within the previous 3 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Overall Patient satisfaction of skin improvement assessed by the Goodman and Barons quantitative scar scale. | 6 months
  A global quantitative grading system for assessing the disease load and global severity of disease in a patient with post acne scarring. The Goodman and Baron score considers type of scar, number of scars, and severity of scarring and assigns a grade 1-4 with grade 1 representing mild, macular disease and grade 4 representing severe scarring that is obviously visible at social distances of 50cm, is not easily covered by makeup, and is not able to be flattened by manual stretching of the skin. Lower scores are favorable. Scale will be completed at every office visit over the 6 month study.
The Global Aesthetic Improvement Scale (GAIS) | 6 months
  The Global Aesthetic Improvement Scale (GAIS) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator 5 point scale ranging from 1 to 5 with 5 = The appearance has worsen compared with the original condition and 1 = Excellent corrective results

SECONDARY OUTCOMES:
Overall Skin changes assessed by Derma Scan | 6 months
  The Derma Scan System utilizes two special lighting systems (RGB +UV) and smart skin analyzer software that allows two images (before and after care) to be compared side by side, which can be used to detect the changes in skin
Overall Skin changes assessed by Acne Scar Subtypes | 6 months
  Skin improvement assessed by Acne Scar Subtypes for improvement of acne scarring rolling, icepick, and or boxcar subtypes.Ice pick scars are narrow, sharply demarcated, V-shaped tracts, <2 mm in diameter, that extend into the deep dermis or even subcutaneous layer. Boxcar scars are wider (1-4 mm in diameter), U-shaped tracts, with sharp, vertical edges that extend 0.1-0.5 mm into the dermis. Rolling scars are characterised by dermal tethering of the dermis to the subcutis. They are generally ≥4 mm in diameter, irregular, with a rolling or undulating appearance.Scale will be completed at every office visit over the 6 month study.
Photographs | 6 months
  Digital imaging device using a grid background with controlled lighting and setting to grade acne scar improvement on a quartile grading scale(1 = 1% to 25%, 2 = 26 to 50%, 3 = 51 to 75%, 4 = >76% improvement).
To evaluate the impact on the quality of life (DLQI) | 6 months
  The Dermatology Life Quality Index questionnaire (DLQI) is 10 questions were asked to the patients and score is 0-3 for each question. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice E Wright, DR, Principal Investigator — Columbia University/ Harlem Hospital HHCNYC; Leslie L Nesbitt, Study Chair — Universal Skincare
Locations (1):
- Lavish Beauty, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once the overall trial is completed and sensitive detailed information is legally advised to published.

REFERENCES:
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Result] Goodman GJ, Baron JA. Postacne scarring: a qualitative global scarring grading system. Dermatol Surg. 2006 Dec;32(12):1458-66. doi: 10.1111/j.1524-4725.2006.32354.x. PMID 17199653
- See also: Derma Scan — http://universalskincareinstitute.com/
- See also: Atrophic Scars Subtypes — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2958495/